CLINICAL TRIAL: NCT01362361
Title: TRICC-C: A Multicenter, Randomized, Phase II Trial: BIBF 1120 vs. Placebo in Patients Receiving Oxaliplatin Plus Fluorouracil and Leucovorin (mFOLFOX6) for Advanced, Chemorefractory Metastatic Colorectal Cancer (mCRC)
Brief Title: TRICC-C (AIO-KRK-0111): BIBF 1120 Versus Placebo in Patients Receiving Oxaliplatin Plus Fluorouracil and Leucovorin (mFOLFOX6) for Advanced, Chemorefractory Metastatic Colorectal Cancer (mCRC)
Acronym: AIO-KRK-0111
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Martin-Luther-Universität Halle-Wittenberg (Other)
Collaborators: GALMED GmbH (Other)
Responsible Party: Principal Investigator, Prof. Dr. med. Thomas Seufferlein, PI, Martin-Luther-Universität Halle-Wittenberg
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TRICC-C (AIO-KRK-0111); 2010-023050-37 (EudraCT Number)
Record Dates: First submitted 2011-05-25; First posted 2011-05-30 (Estimated); Last update posted 2019-09-19 (Actual); Status verified 2019-09

CONDITIONS: Colorectal Cancer
Keywords: Second line colorectal cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — nintedanib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A (Experimental): mFOLFOX6 + BIBF 1120
  Interventions: Drug: mFOLFOX6 + BIBF 1120
- Arm B (Placebo Comparator): mFOLFOX6+placebo
  Interventions: Drug: mFOLFOX6+placebo

INTERVENTIONS:
Drug: mFOLFOX6 + BIBF 1120 — mFOLFOX6 + BIBF1120 (2x200 mg/d d1-d14) (repeated every 14 days)
  Arms: Arm A
Drug: mFOLFOX6+placebo — mFOLFOX6 + placebo (2x200 mg/d d1-d14) (repeated every 14 days)
  Arms: Arm B

SUMMARY:
The purpose of this study:

To explore the comparative effectiveness of BIBF 1120 in terms of :

* Progression-free survival (PFS), objective response, overall survival
* Evaluate and compare safety

ELIGIBILITY:
Inclusion Criteria:

1. Histologically proven colorectal adenocarcinoma
2. Intended treatment with mFOLFOX6 after one prior palliative chemotherapy for metastatic CRC
3. Age > 18 years
4. Metastatic disease not suitable for curative-intent surgery
5. Measurable (> 1 cm) and evaluable disease (according to RECIST 1.1 criteria)
6. Prior bevacizumab, cetuximab or panitumumab are allowed.
7. Previous adjuvant oxaliplatin-containing therapy is allowed, if the end of adjuvant chemotherapy is >12 months prior to inclusion into the trial
8. ECOG performance status 0 or 1 (see appendix 10.4)
9. Adequate hepatic function
10. Adequate Renal function
11. Adequate bone marrow function
12. Other lab parameters: proteinuria < CTCAE grade 2, Prothrombin time and/or partial thromboplastin time < 50 % deviation from normal limits
13. Life expectancy at least 3 months
14. Signed and dated written informed consent prior to admission to the study in accordance with ICH-GCP guidelines and to the local legislation

Exclusion Criteria:

1. Known hypersensitivity to the trial drugs or their excipients.
2. Treatment with any investigational drug within 28 days of trial onset.
3. Prior treatment with more than one line of palliative standard chemotherapy for colorectal cancer, prior treatment with a tyrosine kinase inhibitor, prior palliative treatment with an oxaliplatin-containing regime.
4. History of other malignancies in the last 5 years, in particular those which could affect compliance with the protocol or interpretation of results. Patients with adequately treated basal or squamous cell skin cancer are generally eligible.
5. Serious concomitant disease, especially those that would limit compliance with trial requirements or which are considered relevant for the evaluation of the efficacy or safety of the trial drug, such as neurologic, psychiatric, infectious disease or active ulcers (gastro-intestinal tract, skin) or laboratory abnormality that may increase the risk associated with trial participation or trial drug administration, and in the judgment of the investigator would make the patient inappropriate for entry into the trial.
6. Major injuries and/or surgery or bone fracture within 4 weeks of trial inclusion, or planned surgical procedures during the trial period. Portimplantation prior to therapy is allowed.
7. Significant cardiovascular diseases (i.e. uncontrolled hypertension, unstable angina, history of infarction within past 9 months, congestive heart failure > NYHA II) (see appendix 10.3).
8. History of severe haemorrhagic or thrombotic events in the past 12 months (excluding central venous catheter thrombosis and peripheral deep vein thrombosis). Known inherited predisposition to bleeds or to thrombosis.
9. Patient with brain metastases that are symptomatic and/or require therapy.
10. Therapeutic anticoagulation (except low dose heparin and/or heparin flush as needed for maintenance of an indwelling intravenous device) or antiplatelet therapy (except for chronic low-dose therapy with acetylsalicylic acid ≤ 325mg per day)
11. History of major thrombotic or clinically relevant major bleeding event in the past 6 months
12. Current peripheral neuropathy ≥ CTCAE grade 2 except due to trauma
13. Serious infections requiring systemic antibiotic (e.g antiviral, antimicrobial, antifungal) therapy
14. Gastrointestinal disorders or abnormalities that would interfere with absorption of the study drug
15. Active alcohol or drug abuse.
16. Women and men who are sexually active and unwilling to use a medically acceptable method of contraception
17. Pregnancy or breast-feeding
18. Leptomeningeal disease
19. Radiographic evidence of cavitary or necrotic tumours
20. Centrally located tumours with radiographic evidence (CT or MRI) of local invasion of major blood vessels
21. Severe chemotherapy-associated toxicity during or after adjuvant or palliative first-line chemotherapy like 5-FU-associated cardiac toxicity (coronary spasm) or persistent oxaliplatin-associated peripheral neuropathy (≥ CTCAE grade 2) with paresthesia associated with pain or functional impairment (after adjuvant oxaliplatin-containing chemotherapy).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2011-06; Primary Completion 2016-06 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
progression free survival | 1 year

CONTACTS AND LOCATIONS:
Locations (12):
- Germany (12):
  - Universitätsklinikum Halle, Halle, Saxony-Anhalt
  - Schwerpunktpraxis für Hämatologie und Onkologie Bottrop und Dorsten, Bottrop
  - Kliniken der Stadt Köln gGmbH - Krankenhaus Holweide, Cologne
  - Universitätsklinikum Greifswald -Klinik für Innere Medizin A, Greifswald
  - Gemeinschaftspraxis und Tagesklinik Onkologie und Gastroenterologie - Halle, Halle
  - Klinikum Karlsruhe, Medizinische Klinik III, Karlsruhe
  - Universitätsmedizin Mannheim - TTZ am Interdisziplinären Tumorzentrum, Mannheim
  - Joh. Wesling Klinikum Minden, Minden
  - Stauferklinikum Schwäbisch Gmünd - Mutlangen - Zentrum Innere Medizin, Mutlangen
  - Klinikum der Universität München-Großhadern - Medizinische Klinik und Poliklink III, München
  - Leopoldina-Krankenhaus Schweinfurt - Medizinische Klinik 2, Schweinfurt
  - Universitätsklinikum Ulm - Klinik für Innere Medizin I, Ulm

REFERENCES:
- [Derived] Ettrich TJ, Perkhofer L, Decker T, Hofheinz RD, Heinemann V, Hoffmann T, Hebart HF, Herrmann T, Hannig CV, Buchner-Steudel P, Guthle M, Hermann PC, Berger AW, Seufferlein T. Nintedanib plus mFOLFOX6 as second-line treatment of metastatic, chemorefractory colorectal cancer: The randomised, placebo-controlled, phase II TRICC-C study (AIO-KRK-0111). Int J Cancer. 2021 Mar 15;148(6):1428-1437. doi: 10.1002/ijc.33296. Epub 2020 Oct 4. PMID 32930387